CLINICAL TRIAL: NCT02082301
Title: Oral Glucose Tolerance Testing After Gestational Diabetes
Status: Completed | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Loyola University (Other)
Responsible Party: Principal Investigator, Ted Waters, Principal Investigator, MetroHealth Medical Center
Other Study IDs: IRB12-00581
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Gestational Diabetes; Pregnancy; Obesity
MeSH Terms: conditions — Diabetes, Gestational; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum for measurements of insulin, markers of inflammation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gestational diabetes: Primary cohort is women with diagnosis of gestational diabetes without evidence of overt diabetes

SUMMARY:
This is an observation study of women with gestational diabetes. Subjects recruited undergo immediate postpartum diabetic screening prior to discharge. Post-partum screening for overt diabetes is repeated 6-12 weeks postpartum. The outcome of interest is the utility of an immediate post partum screen for overt diabetes compared to a traditional 6 week test.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational diabetes

Exclusion Criteria:

* Multiple gestations
* pre-pregnancy diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary cohort is obtained from a pregnant population at two academic medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05-04 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Primary outcome: sensitivity of immediate post partum screen | Immediate post partum
  2 hour fasting 75g OGTT immediately post partum. This is compared to a traditional 6 week post partum 75g OGTT for the sensitivity, positive and negative predictive value of the immediate post partum test

SECONDARY OUTCOMES:
Secondary outcome: physiology | 3 time points: antepatum, immediate postpartum, 6 weeks post partum
  A small sub-cohort of women will undergo an additional 2 hour fasting 75g OGTT in the third trimester with measurements of insulin, cytokines, lipids.

CONTACTS AND LOCATIONS:
Overall Officials: Thaddeus Waters, MD, Principal Investigator — Loyola University
Locations (2):
- United States (2):
  - University Hospital, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio

REFERENCES:
- [Derived] Waters TP, Kim SY, Sharma AJ, Schnellinger P, Bobo JK, Woodruff RT, Cubbins LA, Haghiac M, Minium J, Presley L, Wolfe H, Hauguel-de Mouzon S, Adams W, Catalano PM. Longitudinal changes in glucose metabolism in women with gestational diabetes, from late pregnancy to the postpartum period. Diabetologia. 2020 Feb;63(2):385-394. doi: 10.1007/s00125-019-05051-0. Epub 2019 Dec 9. PMID 31820038